CLINICAL TRIAL: NCT04907656
Title: Initial Assessment of the Feasibility and Efficacy of a Scaleable Digital CBT for Generalized Anxiety and Associated Symptoms in a Chronic Musculoskeletal Pain Population
Brief Title: Assessment of the Efficacy of Digital CBT for Anxiety in Adults With Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Principal Investigator, Boston University Charles River Campus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5975E
Record Dates: First submitted 2021-05-18; First posted 2021-06-01 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Pain, Chronic; Pain, Musculoskeletal; Anxiety
Keywords: Anxiety; Worry; Depression; Sleep difficulties; Anxiety sensitivity; Pain intensity; Pain interference
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Anxiety Disorders; Depression; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the dCBT app or a waitlist (control) condition with a 1.5:1 allocation (dCBT:Control) using a blocked randomized sequence. If initially allocated to the control condition, participants will be given access to the dCBT app after week 10 (that is, after the post-treatment evaluation, participants in the control group will be provided (crossed over to) dCBT).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dCBT Condition (Experimental): The dCBT used in this study (Daylight) was selected due to its noted efficacy in treating GAD. 25 interventions will be provided in four modules, with an average duration of 20 minutes. Sessions are unlocked weekly, and completion of an initial assessment drives an algorithm to personalize the program. Individuals may progress through treatment at a slower pace than weekly sessions; 10 weeks is allowed for treatment completion. Treatment is based on principles of applied relaxation, stimulus control, cognitive restructuring, and imaginal exposure. Participants schedule a time for each session and receive prompts if they miss the appointment. All interventions are aided by the use of an animated therapist.
  Interventions: Behavioral: dCBT
- Waitlist (control) Condition (No Intervention): Participants allocated to the waitlist (control) condition will not receive an active intervention during the study. Participants will still complete all scheduled study assessments. They will receive access to the dCBT after completion of all study assessments.

INTERVENTIONS:
Behavioral: dCBT — As per arm of the same name
  Other Names: Daylight
  Arms: dCBT Condition

SUMMARY:
The present study involves a randomized clinical trial of Digital Cognitive Behavioral Therapy (dCBT) targeting worry and anxiety symptoms in a population with chronic pain and clinical levels of generalized anxiety disorder (GAD) symptoms. The clinical trial calls for the recruitment and randomization of 80 individuals with chronic musculoskeletal pain and clinical levels of GAD symptoms to either a dCBT program or a waitlist (Control) condition. The current research represents the first-step investigation of a treatment strategy with the potential to enhance care for patients with chronic pain by introducing a scalable, affordable, and system-friendly digital intervention (dCBT) that targets a prominent source of distress and associated disability in these patients. The investigators propose that by targeting GAD in chronic pain in a way that does not tax engagement in ongoing medical care provision, there is the potential to improve the uptake of effective care and to address both GAD and associated distress and disability.

DETAILED DESCRIPTION:
An emerging body of research points to the significant impact of generalized anxiety disorder (GAD) on the functioning of adults with chronic pain. The importance of managing stress and anxiety is central to the fear/avoidance models of chronic pain, and fears of pain are elevated in those with GAD. Furthermore, the incidence of GAD is significantly higher in patients with chronic pain than in the general population. Likewise, severity of pain, degree of disability, opioid use, and medical costs have been found to be higher among those with comorbid GAD compared to those with chronic pain alone. The treatment of GAD in a chronic pain population has the potential to benefit pain-related distress and disability in addition to direct benefits on GAD and related quality of life.

Cognitive Behavior Therapy (CBT) is an excellent choice for targeting GAD symptoms in a chronic pain population. CBT is a recommended first-line treatment for GAD according to international guidelines. Despite the potential benefits of treatment, individuals with GAD face significant barriers in accessing CBT, including limitations on the availability of trained therapists, the costs and burden of in-person therapy, and stigma issues. These barriers are likely magnified for individuals with chronic pain who also face their own stigma issues as well as a high medical appointment burden. An innovative solution for overcoming these barriers and providing CBT for GAD at scale is to offer well-validated digital treatment that can be delivered by smartphones, tablets, or computers. Digital CBT (dCBT) offers a cost-effective and scalable alternative to in- person CBT with comparable maintenance of treatment gains to in-person CBT at four-year follow-up. Interest in digital health solutions is evident in those with chronic pain, and digital treatment may also offer a strategy for addressing the significant racial and ethnic disparities in care as well as disparities in the degree of psychological distress reported for those with chronic pain. At this time, however, the efficacy of dCBT for GAD has not been evaluated in patients with chronic pain.

The study contains two phases, with only Phase 2 being registered here. Following the achievement of benchmarks from Phase I, Phase 2 is a randomized clinical trial of Digital Cognitive Behavioral Therapy (dCBT) targeting worry and anxiety symptoms in a population with chronic pain and clinical levels of generalized anxiety disorder (GAD) symptoms. The dCBT under study is a commercially available smartphone application that provides weekly intervention sessions in 4 modules. An initial assessment drives an algorithm to personalize the program and individuals will have 10 weeks to complete the treatment. This randomized clinical trial calls for the recruitment and randomization of 80 individuals to either the dCBT program or a waitlist (control) condition. Specific aims for this project are:

1. To show that dCBT leads to lower GAD symptoms relative to the control condition.
2. To evaluate whether dCBT leads to greater changes in the secondary worry, mood, sleep, quality of life, and anxiety sensitivity outcomes than the control condition.
3. To evaluate whether dCBT leads to lower pain distress and disability outcomes than the wait-list control condition.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain patients engaged in noninvasive treatments
* Age 18 or older
* Post acute phase of chronic pain
* Clinical levels of Generalized Anxiety Disorder (GAD) (operationalized by a score of ≥10 on GAD-7)

Exclusion Criteria:

* Factors that may impede the utilization of digital intervention (non-English speaker/literate; no access to a digital device; severely vision impaired, or severe cognitive impairment)
* Pending acute surgery or with a life prognosis of fewer than 6 months
* Current daily opioid use
* The presence [by self-report] of schizophrenia, psychosis, bipolar disorder, seizure disorder, or current substance use disorder (other than nicotine)
* The ability to isolate the effects of the intervention (initiation or change of psychotropic medication dosage within past 4 weeks, received CBT for anxiety in last 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Anxiety Severity | Week 10
  The Generalized Anxiety Disorder 7 (GAD 7) is a self-report measure that assesses the full range of symptoms associated with GAD. Responses are summed to create a composite score, with higher scores indicating more severe anxiety. Composite scores range from 0 to 21.

SECONDARY OUTCOMES:
Worry Severity | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Penn State Worry Questionnaire (PSWQ) is a self report measure of worry. Responses are summed to create a composite score, with higher scores indicating more severe worry. Composite scores range from 16 to 80.
Depression | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Patient Health Questionnaire (PHQ-8) is a self report measure of depression symptoms experienced in the past two weeks. It excludes the suicide item of the PHQ-9.
Sleep Difficulty | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Sleep Condition Indicator (SCI) is a self-report measure used to assess sleep related difficulties and insomnia based on the DSM-5 criteria. All 8 items are summed to create the composite score. Possible composite scores range from 0 to 32, with higher scores indicating better sleep.
Health status | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Short Form Health Survey (SF-12) is a self-report measure that assesses quality of life related to both physical and mental health. This measure does not have public scoring details and uses a weighted scoring algorithm. The average of select items is computed for subscale scores (physical and mental). Scores range from 0 to 100, with higher scores indicating better health/well-being and no disability.
Anxiety sensitivity | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Anxiety Sensitivity Index (ASI-3) is a self-report measure that assess three dimensions of anxiety sensitivity: fear of physical symptoms, fear of cognitive dyscontrol, and fear of social concerns. All 18 items are summed to create the composite score, with higher scores indicating more severe anxiety sensitivity.
Clinician-rated anxiety severity | Week 0 (baseline), Week 10 (post-intervention)
  The Hamilton Anxiety Rating Scale (HARS) will be administered per the structured interview guide for this instrument to provide a clinician-rated measure of anxiety severity. Detailed scoring instructions are available in the interview guide; composite scores range from 0 to 56, with higher scores indicating more severe distress and impairment.
Pain intensity | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Brief Pain Inventory (BPI) is a self-report measure with 4 items used to assess pain severity. The severity score is the mean of the 4 items. Scores can range from 0 to 10, with higher scores indicating more intense pain.
Pain interference/disability | Week 0 (baseline), week 6, week 10 (post-intervention)
  The BPI is a self-report measure with 7 items used to assess pain disability/interference. The interference score is the mean of the 7 items. The mean can be used if 50%, or 4 of the 7, items are completed. Scores can range from 0 to 10, with higher scores indicating more complete interference.
Fear of pain | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Pain Anxiety Symptoms Scale (PASS-20) is a self-report used to assess fear of pain. Responses are summed to create a composite score, ranging from 0 to 100 with higher scores indicating more severe fear of pain
Pain medication use | Week 0 (baseline), week 6, week 10 (post-intervention)
  Use of pain medication and other pain interventions will be assessed with a self-report form developed by the research team for use in this study. Based on a composite scoring of medication dosages reported by participants, pain medication use at week 6 and week 10 will be coded as an increase, decrease, or steady state from the baseline dosages.
Pain catastrophizing | Week 0 (baseline), week 6, week 10 (post-intervention)
  The Pain Catastrophizing Scale (PCS) is a self-report measure used to assess catastrophic thinking related to pain. Responses to all 13 items are summed to create a composite score, with higher scores indicating more severe catastrophic thinking. Scores range from 0 to 52.
Anxiety Severity | Week 0 (baseline), week 3, week 6
  The Generalized Anxiety Disorder 7 (GAD 7) is a self-report measure that assesses the full range of symptoms associated with GAD. Responses are summed to create a composite score, with higher scores indicating more severe anxiety. Composite scores range from 0 to 21.
Resolution of clinical GAD | Week 10 (post-intervention)
  The proportion of participants no longer meeting GAD-7 clinical severity, operationalized as a score of less than 10 at the week 10 evaluation. Scoring will be the same as described for the GAD-7 above.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Otto, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States